CLINICAL TRIAL: NCT05032781
Title: Intra-Arterial Administration of Neuroprotective Agents and Cold Saline at Time of Recanalization for Acute Ischemic Stroke Due to Large Vessel Occlusion
Brief Title: Intra-Arterial Neuroprotective Agents and Cold Saline in Ischemic Stroke Intervention
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-1198
Record Dates: First submitted 2021-05-04; First posted 2021-09-02 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Ischemic
Keywords: Ischemic stroke; Large vessel occlusion; Mechanical thrombectomy; Neuroprotection; cold saline; Minocycline; Magnesium sulfate
MeSH Terms: conditions — Ischemic Stroke; cyclopia sequence | interventions — Minocycline; Magnesium

STUDY DESIGN:
Intervention Model Description: See study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intra-arterial neuroprotective substances (Experimental): Cold saline, minocycline, and magnesium sulfate to be infused intra-arterially immediately after thrombectomy via the internal carotid artery. A dose escalation design will be used, as described above in "Study Description."
  Interventions: Drug: Intra-arterial cold saline, minocycline, and magnesium

INTERVENTIONS:
Drug: Intra-arterial cold saline, minocycline, and magnesium — See study design

SUMMARY:
Ischemic stroke is the leading cause of long-term disability in the United States. Endovascular intervention with mechanical thrombectomy has become the standard of care for acute large vessel occlusion (LVO) stroke since multiple clinical trials demonstrated improved long-term clinical outcomes with treatment. However, despite high rates of successful vessel recanalization and thus reperfusion of ischemic brain tissue in current practice, many patients continue to suffer debilitating strokes and poor long-term functional outcome. Pharmacologic neuroprotection could potentially present a means of addressing this mismatch in radiologic vs. clinical outcomes by protecting and salvaging damaged brain tissue. Intra-arterial delivery of a cocktail of neuroprotective therapy at the time of endovascular reperfusion would provide immediate, targeted therapy directly to the damaged brain territory. Hypothermia, minocycline and magnesium can target multiple facets of the complex ischemic injury cascade, and have each demonstrated neuroprotection in multiple preclinical models. This is a phase I trial that aims to demonstrate safety and feasibility of administering cold saline, minocycline, and magnesium sulfate intra-arterially immediately after thrombectomy in stroke interventions.

DETAILED DESCRIPTION:
This is a phase I, single center, single arm clinical trial with dose escalation design.

Location: North Shore University Hospital in Manhasset, NY

Study population: Subjects aged 18-90 years undergoing mechanical thrombectomy for acute ischemic stroke due to large vessel occlusion at North Shore University Hospital

Primary Objective: To demonstrate the safety and feasibility of intra-arterial administration of a cocktail of neuroprotective agents at the time of reperfusion in endovascular stroke intervention for acute ischemic stroke due to large vessel occlusion.

Secondary Objectives:

A) To describe the feasibility of delivering a combination of neuroprotective agents directly into the affected internal carotid artery immediately after recanalization of an occluded vessel in ischemic stroke intervention.

B) To describe the maximum tolerated dose of a combination of 4C saline at 30 ml/min for 10 minutes, minocycline, and magnesium sulfate directly into the affected internal carotid artery immediately after recanalization of an occluded vessel in ischemic stroke intervention.

C) To describe the clinical outcomes of the patients undergoing the experimental procedure and compare to historical controls.

Primary Endpoint: Presence of symptomatic intracranial hemorrhage within 24 hours of treatment; presence of serious adverse event related to the administration of intra-arterial cold saline, minocycline or MgSO4; and technical feasibility of the proposed experimental treatment.

Secondary Endpoints: Total volume of infarct on MRI 24 hours after procedure, clinical outcome as measured by the NIHSS prior to discharge and MRS at 90 day follow up.

Study design:

Based on the available literature, the target dose of Minocycline and MgSO4 is 6 mg/kg and 2g, respectively. For targeted hypothermia, 4C normal saline will be infused at a rate of 30 ml/min to achieve an estimated drop in temperature in the ipsilateral hemisphere to 33-34C within 10 minutes.

To ensure adequate safety measures, a dose escalation design is employed to carefully evaluate for adverse events throughout the study. The standard "3+3" dose escalation design will be used in the 3 groups described below. Within each group, at each dosage, if none of the first 3 patients experience a related adverse event, the study proceeds to the next group or dose level. If one of the 3 patients experiences an adverse event, then an additional 3 patients will be treated at that dose level before proceeding. Escalation will continue only if a maximum of 1 out of 6 patients experience an adverse event. If 2 or more patients at a given dose level experience an adverse event, then the maximum tolerated dose (MTD) will be determined as the preceding dose level.

Group 1: IA cold saline alone 3-6 patients receive 4C at 30 ml/min over 10 min

Group 2: IA cold saline + Minocycline 3-6 patients receive IA cold saline + 2 mg/kg Minocycline; 3-6 patients receive IA cold saline + 4 mg/kg Minocycline; 3-6 patients receive IA cold saline + 6 mg/kg Minocycline

Group 3: IA cold saline + Minocycline + Magnesium sulfate 3-6 patients receive IA cold saline + MTD Minocycline + 2g MgSO4; 3-6 patients receive IA cold saline + MTD Minocycline + 4g MgSO4

Both the Minocycline and MgSO4 will be reconstituted within the 300 ml of cold saline to be administered together.

Follow up:

Post-stroke intervention care will proceed as standard of care with the addition of screening for adverse events related to the IA administration of cold saline, minocycline and/or magnesium sulfate.

Day 1: CT or MRI within 24h of intervention, neurologic exam, routine labs, NIHSS.

Day of discharge: neurologic exam, routine labs, NIHSS, mRS. Day 90: neurologic exam, NIHSS, mRS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-90
* Signed and dated informed consent and IRB form by the patient or legally authorized health care proxy.
* Diagnosis of acute ischemic stroke due to large vessel occlusion based on clinical and radiographic evidence as determined and documented by the Stroke Neurology team at Northshore University Hospital.
* Participants must meet criteria for intra-arterial thrombectomy as determined and documented by the Stroke Neurology and Interventional Neuroradiology attending physicians at Northshore University Hospital.
* Angiography must reveal a thromboembolism which is completely occluding flow within the intracranial portion of the internal carotid artery, the M1 or proximal M2 portions of the middle cerebral artery.

Exclusion Criteria:

* Patients that do not otherwise meet criteria for endovascular intervention
* Large vessel occlusion of the anterior cerebral artery, posterior circulation, or distal M2 portion of the middle cerebral artery.
* Recanalization of only TICI 0-2A.
* Pregnant or lactating women.
* Therapeutic anticoagulation prior to presentation.
* Known allergic reactions to contrast dye or components of minocycline (tetracycline) or magnesium sulfate.
* Patients with a known prior diagnosis of heart block or prior myocardial infarction (increased risk of adverse reaction to MgSO4).
* Renal insufficiency (creatinine > 2.5 mg/dL)
* Severe hepatic functional impairment (AST > 10xULN, bilirubin > 5xULN)
* Systemic lupus erythematosus
* Idiopathic intracranial hypertension

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Intracranial hemorrhage | within 24 hours of treatment
  Presence of symptomatic intracranial hemorrhage
Presence of serious adverse event | within 72 hours of treatment
  Related to intra-arterial administration of cold saline, minocycline, or magnesium sulfate

SECONDARY OUTCOMES:
Infarct volume | 24 hours after procedure
  Total volume of infarct on MRI
Functional outcome | 90 days after intervention
  Clinical outcome as determined by modified Rankin scale (0-6)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Link, MD, MS, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No